CLINICAL TRIAL: NCT02062723
Title: Prospective Observational Study to Assess the Efficacy and Tolerability of Eptadone®, in Heroin Addicted Patients Undergoing a Methadone Maintenance Treatment
Brief Title: Observational Study to Assess the Efficacy and Tolerability of Eptadone®, in Heroin Addicted Patients in a MMT
Acronym: METHODE
Status: Completed | Type: Observational
Sponsor: L.Molteni & C. dei F.lli Alitti-Soc. di Esercizio S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: MOLT-2009-002
Record Dates: First submitted 2014-01-24; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Heroin Addiction
Keywords: methadone; heroin addiction; methadone maintenance treatment; adequate dosage of methadone
MeSH Terms: conditions — Heroin Dependence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pts addicted to heroin in MMT: patients addicted to heroin who have undertaken methadone maintenance treatment

SUMMARY:
The efficacy and tolerability of Eptadone® in the context of a maintenance program will be evaluated in an observational prospective, multicenter study, in heroin addicted patients.

DETAILED DESCRIPTION:
515 patients have been selected among all patients addicted to heroin according ICD-10, in maintenance treatment with Eptadone, observed in the involved sites. The investigators have used the treatment schemes with Eptadone conform to the registered use.

The enrollment has been competitive. Patients met incl/excl and that have signed the informed consent have been observed for 1 year. Follow up visits have been performed according to routine procedures, for patients related to the centres at 3/6/12 months post V1. During the visits patients have been assessed by validated and used as clinical practice questionaries. Safety and tolerability have been assessed through the collection of adverse reactions and of laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Over 18 years of age
* Patients with a diagnosis of heroin addiction, according to ICD-10 (International Classification of Diseases-10)
* Patients who receive a "maintenance treatment" with Eptadone® since at least one month
* Accession to the observational study by informed consent

Exclusion Criteria:

* Inability to follow the observation and to understand study procedure and follow them
* Diagnosis of:

  * Decompensated psychotic disorders,
  * Epileptic attacks, not related with drug abuse,
  * Severe-acute or severe-chronic somatic diseases (like AIDS, Tubercolosis, acute hepatitis, Sepsis ecc), whereas chronical HCV is not an exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with heroin addiction, over 18 years of age.
Sampling Method: Probability Sample
Enrollment: 515 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Primary endpoint | From baseline to end of study (12 months after baseline)
  Efficacy and Tolerability of maintenance treatment with Eptadone®, in patients addicted to heroin.

SECONDARY OUTCOMES:
Secondary endpoints | From baseline to end of study (12 months after baseline)
  Pharmacoeconomic evaluation of the maintenance treatment with Eptadone®; compliance of patients to the treatment with Eptadone®; efficacy of Eptadone® in relation to sex and group of age; effects of methadone on sexual functioning.

CONTACTS AND LOCATIONS:
Locations (22):
- Germany (22):
  - Facharzt für Allgemeinmedizin, Bad Honnef
  - Praxis Turmstrasse, Berlin
  - Praktischer Arzt, Bonn
  - Arzt für Allgemeinmedizin, Bremen
  - Psychiatrie, Bremen
  - Praxis, Cologne
  - Dres. Beck & Hummel Artzegemeinschaft, Fürstenfeldbruck
  - Gemeinschaftspraxis fur Neurologie, Psychiatrie und Suchtmedizin Poliklinik Silberhohe, Halle
  - Universitätsklinikum Hamburg-Eppendorf Klinik und Poliklinik fur Psychiatrie und Psychotherapie, Hamburg
  - Arzt für Allgemeinmedizin, Hamburg
  - Gemeinschaftspraxis Suchtmedizin, Hamburg
  - Fachgebiet Allgemeinmedizin, Hamburg
  - Praxiszentrum Friedrichsplatz, Kassel
  - Facharzt für Psychiatrie Psychotherapie, Lehrte
  - Facharzt für Innere Medizin, Leipzig
  - Praxiszentrum im Tal, München
  - Praxis, München
  - Concept Schwerpunktpraxis Sucht, München
  - Facharzt fur Psychiatrie, Münster
  - Hausärztliche Praxis, Regensburg
  - Bezirksklinik Regensburg, Regensburg
  - Psychatrie, Ulm